CLINICAL TRIAL: NCT01197157
Title: Impact of Nitazoxanide on Virologic Responses in Chronic HCV Infected Patients With Genotype 4: A Placebo-controlled Randomized Trial
Brief Title: Study of the Impact of Nitazoxanide on Chronic Hepatitis Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Liver Institute, Egypt (Other)
Responsible Party: Principal Investigator, Mohamed Kohla, Lecturer of Hepatology, National Liver Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NEAR trial
Record Dates: First submitted 2010-08-09; First posted 2010-09-09 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Hepatitis C
Keywords: chronic hepatitis C; genotype 4; treatment naive patients; Egypt
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — Control Groups; nitazoxanide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): • Group A: comprises 100 chronic hepatitis patients who will receive placebo twice daily orally with food for an average of 12 weeks followed by the standard of care treatment, peginterferon Alfa 2a once weekly and weight-based ribavirin 1000 or 1200 mg/day (based on body weight < 75 kg or ≥ 75 kg, respectively) in divided doses plus placebo twice daily for 48 weeks.
  All patients in this group will have an HCV RNA within 3 months before initiation of therapy, in addition to ALT levels, CBC and other routine liver function tests.
  Interventions: Drug: Placebo
- Nitazoxanide (Experimental): • Group B: comprises 100 CHC patients who will receive oral Nitazoxanide 500 mg twice daily with food for an average of 12 weeks as a part of monotherapy lead-in phase followed by triple therapy, nitazoxanide 500 mg twice daily plus peginterferon alfa-2a (once weekly), and weight-based ribavirin (1000-1200 mg daily) for 48 weeks.
  All patients in this group will have an HCV RNA within 3 months before initiation of therapy, in addition to ALT levels, CBC and other routine liver function tests.
  Interventions: Drug: Nitazoxanide

INTERVENTIONS:
Drug: Placebo — Group A: comprises 100 CHC patients who will receive placebo twice daily with food for an average of 12 weeks as a part of monotherapy lead-in phase followed by triple therapy, nitazoxanide 500 mg twice daily plus peginterferon alfa-2a (once weekly), and weight-based ribavirin (1000-1200 mg daily) for 48 weeks.
  Other Names: Control group
  Arms: placebo
Drug: Nitazoxanide — • Group B: comprises 100 chronic hepatitis patients who will receive oral Nitazoxanide 500 mg twice daily with food for an average of 12 weeks followed by the standard of care treatment, peginterferon Alfa 2a once weekly and weight-based ribavirin 1000 or 1200 mg/day (based on body weight < 75 kg or ≥ 75 kg, respectively) in divided doses plus placebo twice daily for 48 weeks.
  Other Names: Alinia; Xerovirinc(Minapharm Pharmaceuticals)
  Arms: Nitazoxanide

SUMMARY:
The main objective of antiviral therapy of patients with chronic hepatitis C (CHC) is the sustained elimination of the hepatitis C virus (HCV). The standard of care (SOC) is peginterferon alfa-2a/-2b with ribavirin for 48 weeks or 24 weeks according to HCV genotype.

However, this approach is not sufficient to substantially improve the sustained virologic response (SVR) rates. Therefore, new therapies are needed to treat patients with hepatitis C virus (HCV) infection. Nitazoxanide (NTZ), originally used to treat cryptosporidium parvum infection, recently was shown to have an unexpected antiviral activity in the HCV replicon system and in chronically infected patients.

The aim of this work is to study impact of nitazoxanide therapy in addition to peginterferon/ribavirin combination on virologic responses in patients with chronic hepatitis C genotype 4.

Patients will be enrolled in this study and will be randomly assigned in a 1:1 ratio into 2 groups:

Group A: comprises 100 CHC patients who will receive the standard of care treatment, peginterferon-alf 2a plus weight-based ribavirin for 48 weeks.

Group B: comprises 100 CHC patients who will receive nitazoxanide monotherapy at a dose of 500 mg twice daily for 12 weeks as a lead-in phase followed by triple therapy, nitazoxanide 500 mg twice daily plus peginterferon alfa-2a, and weight-based ribavirin for 48 weeks.

Data will be collected and statistical analysis will be done comparing the groups regarding response to antiviral therapy. Final results will be discussed and compared to similar studies published in peer reviewed journals and international conferences.

DETAILED DESCRIPTION:
Chronic hepatitis C virus (CHC) infects approximately 170 million individuals worldwide. Egypt has the highest hepatitis C virus prevalence in the world (overall prevalence is 12% among the general population, and up to 40% in persons above 40 years of age and is more in rural areas.

Approximately, 90% of hepatitis C patients in Egypt are infected with HCV genotype 4.

The main objective of antiviral therapy of patients with chronic hepatitis C is the sustained elimination of the hepatitis C virus (HCV).

The standard of care for the treatment of chronic hepatitis C is a 24- to 48- week course of peginterferon plus ribavirin, depending on genotype.

Overall, approximately, half of the patients can be cured by SOC. For patients with genotype 4, the sustained virologic response (SVR) rate with 48 weeks of therapy ranges from 50 to 60 %. Based on baseline viral load and the speed of virologic response during treatment, individualization of treatment duration is possible. However, this approach is not sufficient to substantially improve the sustained virologic response (SVR) rates. A significant proportion of treated patients thus either fail to respond or relapse following an initial response and a substantial number of patients are unable to tolerate treatment. There is at present no alternative therapy for these patients and thus a need for new drugs for the treatment of chronic hepatitis C.

Nitazoxanide, the first member of the thiazolidide anti-infective class of compounds, is an oral anti-parasitic agent with no major side effects that was developed and licensed in the US (Alinia; Romark Laboratories, L.C., Tampa FL, USA) for the treatment of cryptosporidium parvum and Giardia lamblia, recently was shown to have an unexpected antiviral activity in the HCV replicon system and in chronically infected patients. A serendipitous observation during drug development revealed that some patients with cryptosporidiosis and acquired immunodeficiency syndrome who are co-infected with hepatitis C or B viruses, had a reduction in serum alanine aminotransferase (ALT) levels during therapy. This observation led to studies of the anti-viral activity of nitazoxanide and its active metabolite tizoxanide in HCV genotype 1a and 1b replicons and a genotype 2 infectious clone, which showed a potent inhibition of HCV replication by both compounds at submicromolar concentrations.

In addition, pretreatment of HCV replicon-containing cells with nitazoxanide was shown to enhance the antiviral effect of subsequent treatment with nitazoxanide plus interferon.

The mechanism of action of nitazoxanide in protozoa and anaerobic bacteria has been shown to result from direct inhibition of pyruvate ferredoxin oxidoreductase enzyme-dependent electron transfer reaction which is essential to anaerobic energy metabolism. However, the antiviral mechanism of action of nitazoxanide appears to be different.

Recent studies of the mechanism of action of nitazoxanide against HCV have shown that it induces double-stranded RNA-activated protein kinase (PKR) phosphorylation, which results in an increased intracellular concentration of phosphorylated eukaryotic initiation factor 2α, a naturally occurring antiviral intracellular protein and a key mediator of host cell defenses against viral infection, this mechanism of action is triggered only when a cell is infected with HCV, whereas nitazoxanide has no effect on in uninfected cells, which provides a potential explanation for its very low rate of toxicity.

It worth mentioning that resistance to nitazoxanide is unlikely as it exerts its antiviral activity by modulating cell signaling, an interferon-like mechanism, rather than by targeting the virus directly and that nitazoxanide does not induce mutations that confer viral resistance, suggesting that the genetic barrier to the development of resistance to nitazoxanide is high.

These clinical and laboratory observations prompted study of the potential effect of nitazoxanide in patients with chronic hepatitis C.

Rossingol JF et al,demonstrated that treatment with nitazoxanide monotherapy at a dose of 500 mg twice daily orally, was associated with an ETR in 7 of 23 (30.4%) patients with chronic hepatitis C genotype 4, the virologic responses occurred between 4 and 20 weeks of therapy (three at week 4, three at week 8 and one at week 20) and continued through the end of treatment with no virological breakthroughs. A low serum HCV RNA ≤ 400,000 IU/ml, was the most significant predictor of virological response (p=0.009). In addition, none of the patients with cirrhosis, poorly controlled diabetes, or the one patient with HBV coinfection responded to treatment. Four of the 7 patients with an ETR (17.4% of 23 treated patients) had an SVR, 24 weeks after the end of treatment.

This preliminary data prompted the study of the efficacy and safety of Nitazoxanide as a triple therapy in combination with peginterferon and ribavirin in patients with chronic hepatitis C genotype 4 aiming at improving the rate of sustained virological response (SVR).

A recent study by Rossignol JF et al, conducted on a total 97 treatment -naïve patients conducted in 2 centers in Egypt demonstrated that, significantly more patients receiving triple therapy with peginterferon alfa-2a, ribavirin and nitazoxanide experienced SVR compared with the standard of care (79% vs 50%; p=0-023). The SVR rates for the peginterferon plus nitazoxanide group was higher than the standard of care (61% vs 50%) although this difference was not statistically significant.

The percentages of rapid virologic response (RVR), defined as undetectable HCV RNA at week 4 of combination therapy, and SVR were significantly higher in patients given the triple (Nitazoxanide/ peginterferon/ ribavirin) therapy compared with the standard of care (64% vs 38%, P = .048; and 79% vs 50%, P = .023; respectively). Patients given nitazoxanide plus peginterferon alfa-2a had intermediate rates of RVR (54%). There were no added side effects associated with the use of nitazoxanide.

Mean reductions in serum HCV RNA from baseline to the RVR visit were -2.86, -3.74, and -4.5 log10 IU/ml for the peginterferon plus ribavirin, dual therapy with peginterferon plus nitazoxanide, and triple therapy with peginterferon, ribavirin and nitazoxanide groups, respectively (p=0.008).

Changes in ALT levels from baseline to week 72 in patients who achieved an SVR were evaluated, nearly all patients had normalization of ALT levels (15/16 patients in groups 1 and 3, and all patients in group 2), in parallel with loss of detectable serum HCV RNA. Interestingly, the use of nitazoxanide in the dual- and triple-treatment arms was associated with reduced relapse rates (3/20 patients and 1/23 patients, respectively) compared with the standard of care arm (10/30 patients).

The rationale for a nitazoxanide lead-in phase before combined therapy with peginterferon, with or without ribavirin, was based on an initial pilot experience that showed greater antiviral efficacy if nitazoxanide was administered before peginterferon rather than simultaneously.

The required duration of nitazoxanide lead-in phase is unknown, and 12 weeks was selected as an initial conservative estimate to optimize the potential benefit of nitazoxanide pretreatment. A subsequent study has shown that a 4-week lead-in phase may be satisfactory, and this study also provides further confirmation of the antiviral efficacy of nitazoxanide combined with peginterferon.

In this open-labeled study, 44 treatment-naïve patients with chronic hepatitis C were treated with 4 weeks on nitazoxanide 500 mg twice daily followed by combination dual therapy of peginterferon alfa-2a 180 µg weekly plus nitazoxanide 500 mg twice daily for an additional 36 weeks. Interestingly, the SVR rate with dual therapy (80%), was similar to the SVR rate with triple therapy (79%) seen in the previous study using a 12-week lead-in phase. This shorter lead-in period might be adequate.

In a preliminary experience with interferon nonresponders, a small number of patients with chronic hepatitis C genotype 4 who had failed prior interferon-based therapy were re-treated using triple therapy with nitazoxanide, peginterferon and ribavirin and achieved an SVR rate of 25% (3/12 patients) compared with 8% (1/12 patients) retreated with the standard of care using peginterferon alfa-2a plus ribavirin.

All these data show that nitazoxanide, a novel protein kinase inducer, has the potential to increase the SVR rate in patients with chronic hepatitis C, however, further studies to test these hypotheses on larger numbers of both naïve and nonresponder patients are still required.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and <60.
* Liver biopsy showing chronic hepatitis with significant fibrosis using Ishak scoring system.
* Compensated liver disease; serum bilirubin < 1.5 mg/dl, INR no more than 1.5, serum albumin > 3.4, platelet count >75,000 mm, and no evidence of hepatic decompensation (hepatic encephalopathy or ascites).
* Acceptable hematological and biochemical indices (hemoglobin 13g/dl for men and 12 g/dl for women; neutrophil count 1500/mm3 or more and serum creatinine <1.5 mg/dl.
* Willing to be treated and to adhere to treatment requirements

Exclusion Criteria:

* Major uncontrolled depressive illness.
* Solid organ transplantation.
* Autoimmune conditions, known to be exacerbated by peginterferon and ribavirin.
* Untreated thyroid disease.
* Pregnant or unwilling to comply with adequate contraception.
* Severe concurrent medical disease such as severe hypertension, heart failure, significant coronary heart disease, poorly controlled diabetes, chronic obstructive pulmonary disease.
* Known hypersensitivity to drugs used to treat HCV.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2010-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Assessment of efficacy of Nitazoxanide as an add-on therapy in terms of achieving a sustained virologic response | 180 ± 7 days after the end of triple therapy, the preliminary data will be available at least 2 years after the beginning of the study (September 2012)
  Patients in the 2 group who will continue on triple therapy till achieving an end-of-treatment response (after 48 weeks from the start of triple therapy), will have their viral load measured 6 months thereafter for assessment of sustained virologic response. patients in whom the virus is undetectble will be regarded as achieving a sustained virologic response.

SECONDARY OUTCOMES:
assessment of rapid virologic response | 28-35 days from the start of triple therapy
  Patients in the 2 groups will have their viral load measured at 4 weeks from the start of triple therapy which is a strong predictor of attaining a sustained virologic response. patients in whom the virus is undetectable will be regarded as achieving a rapid virologic response.
Assessment of early virologic response | 90 ± 7 days from the start of triple therapy
  Patients in the 2 groups will have their viral load measured at 12 weeks from the start of triple therapy. Patients in whom the virus is undetectable, will be regarded as achieving an early virologic response.
Assessment of end-of-treatment response | 48± one week from the start of triple therapy
  Patients in the 2 groups will have their viral load measured at the end of triple therapy (48 weeks). Patients in whom the virus is undetectable, will be regarded as achieving an end-of-treatment response.
Safety of Nitazoxanide | Throughout the study and up to 90 days after the end of triple therapy
  Safety of nitazoxanide will be assesses and all adverse events will be reported, and treatment will be discontinued if necessary
Assessment of the efficacy of Nitazoxanide monotherapy following the lead-in phase | 90± 7 days from the start of the lead_in phase
  Patients in the 2 groups will have their viral load as well as transaminases (ALT&AST) measured at the end of the lead-in phase. in case of a reduction in viral load, this will be expressed as log10 reduction from nadir, also, reduction in serum transaminases from pre-treatment values will be regarded as achieving a biochemical response.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Kohla, MD, Principal Investigator — National Liver Institute, Menoufiya University, Egypt; Hossam A Taha, MD, Study Director — National Liver Institute, Menoufiya University, Egypt
Locations (1):
- National Liver Institute, Shebin El-Kom, Monufia Governorate, Egypt